CLINICAL TRIAL: NCT03610724
Title: A Phase II, Single Arm, Multicenter Open Label Trial to Determine the Safety and Efficacy of Tisagenlecleucel in Pediatric Subjects With Relapsed or Refractory Mature B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Phase II Open Label Trial to Determine Safety & Efficacy of Tisagenlecleucel in Pediatric Non-Hodgkin Lymphoma Patients
Acronym: BIANCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019C2202; 2017-005019-15 (EudraCT Number)
Record Dates: First submitted 2018-07-13; First posted 2018-08-01 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Tisagenlecleucel; CTL019; r/r; relapsed/refractory B-cell non-Hodgkin lymphoma; r/r B-cell NHL subject population; B-cell NHL including Burkitt lymphoma and Burkitt Leukemia; pediatric patients; adolescents; young adults; Burkitt lymphoma (BL); Burkitt leukemia (BL); diffuse large B-cell lymphoma (DLBCL); primary mediastinal large B-cell lymphoma (PMBCL); gray zone lymphoma (GZL); follicular lymphoma (FL); leukapheresis; lymphodepleting chemotherapy (LD); non-Hodgkin lymphoma; NHL; r/r B-NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — tisagenlecleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tisagenlecleucel (Experimental): Participants were infused once with CAR-positive viable T cells
  Interventions: Biological: Tisagenlecleucel; Drug: lymphodepleting chemotherapy; Drug: Bridging Therapy

INTERVENTIONS:
Biological: Tisagenlecleucel — Tisagenlecleucel was infused once as an intravenous infustion at a dose of either 0.2 to 5 x 106 CAR-positive viable T cells per kg body weight for subjects ≤ 50 kg or 0.1 to 2.5 x 108 CAR-positive viable T cells for subjects > 50 kg.
  Other Names: CTL019
Drug: lymphodepleting chemotherapy — Prior to tisagenlecleucel infusion, each subject underwent lymphodepletion with recommended Fludarabine and cyclophosphamide (unless contra-indicated for subject)
Drug: Bridging Therapy — Pre-treatment phase could also include bridging therapy of investigator's choice

SUMMARY:
The purpose of the study was to assess the efficacy and safety of tisagenlecleucel in pediatric, adolescent and young adult patients with relapsed/refractory B-cell non-Hodgkin lymphoma (r/r B-NHL) including Burkitt Lymphoma and Burkitt Leukemia.

For pediatric patients who have r/r B-NHL including Burkitt Lymphoma and Burkitt Leukemia, survival rates are dismal, only ~20-50% subjects are alive at 2 years with overall response rate (ORR) of 20-30% after conventional salvage chemotherapy.

DETAILED DESCRIPTION:
This study was part of an agreed Pediatric Investigation Plan (PIP). The single-arm study design included r/r B-cell NHL including Burkitt Lymphoma and Burkitt Leukemia subject population with poor prognosis, lack of approved effective therapies in this setting. Subject population included aggressive subtypes of B-cell NHL including Burkitt Lymphoma and Burkitt Leukemia who were allowed to receive "bridging therapy" of investigator's choice. After assessment of eligibility, subjects qualifying for the study were enrolled and were allowed to start lymphodepleting chemotherapy as recommended in protocol after which a single dose of tisagenlecleucel product was infused. The efficacy of tisagenlecleucel was evaluated through the primary endpoint of Overall Response Rate (ORR) which included complete response (CR) and partial response (PR) as determined by local assessment. Safety assessments were conducted until study completion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pediatric mature B-cell non-Hodgkin lymphoma (B-cell NHL) including the following subtypes; Burkitt lymphoma/ Burkitt leukemia (BL), diffuse large B-cell lymphoma (DLBCL), primary mediastinal B-cell lymphoma (PMBCL), gray zone lymphoma (GZL), and follicular lymphoma (FL) Note: Patients with B-cell NHL associated with Nijmegen breakage syndrome will be allowed.
* Patients <25 years of age and weighing at least 6 kg at the time of screening
* Patients who have relapsed after one or more prior therapies (can include allogeneic and autologous hematopoietic stem cell transplant) or are primary refractory (have not achieved a CR or PR after the first line of therapy)
* Measurable disease by radiological criteria in all patients at the time of screening. Patients with Burkitt leukemia who don't meet radiological criteria must have bone marrow involvement of >25% by local assessment of bone marrow aspirate and/or biopsy.
* Karnofsky (age ≥16 years) or Lansky (age <16 years) performance status ≥60.
* Adequate bone marrow reserve without transfusions (transfusion >2 weeks prior to laboratory assessment is allowed) defined as:

  1. Absolute neutrophil count (ANC) >1000/mm3
  2. Platelets ≥50000//mm3
  3. Hemoglobin ≥8.0 g/dl
* Adequate organ function defined as:

  1. a serum creatinine (sCR) based on gender/age as follows: Maximum Serum Creatinine (mg/dL) Age Male Female

     1 to <2 years 0.6 0.6 2 to <6 years 0.8 0.8 6 to <10 years 1.0 1.0 10 to <13 years 1.2 1.2 13 to <16 years 1.5 1.4

     ≥16 years 1.7 1.4
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5 times the upper limit of normal (ULN) for age
  3. Total bilirubin <2 mg/dL (for Gilbert's Syndrome patients total bilirubin <4 mg/dL)
  4. Adequate pulmonary function

  i. Oxygen saturation of >91% on room air ii. No or mild dyspnea (≤Grade 1)
* Must have a leukapheresis material of non-mobilized cells accepted for manufacturing.

Exclusion Criteria:

* Prior gene therapy or engineered T cell therapy.
* Prior treatment with any anti-CD19 therapy.
* Allogeneic hematopoietic stem cell transplant (HSCT) <3 months prior to screening and ≤4 months prior to infusion.
* Presence of grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD) in patients who received prior allogeneic HSCT.
* Prior diagnosis of malignancy other than study indication, and not disease free for 5 years.
* Clinically significant active infection confirmed by clinical evidence, imaging, or positive laboratory tests (e.g., blood cultures, PCR for DNA/RNA, etc.)
* Presence of active hepatitis B or C as indicated by serology.
* Human Immunodeficiency Virus (HIV) positive test.
* Active neurological autoimmune or inflammatory disorders not related to B cell NHL (eg: Guillain-Barre syndrome, Amyotrophic Lateral Sclerosis)
* Active central nervous system (CNS) involvement by malignancy.
* Patients with B-cell NHL in the context of post-transplant lymphoproliferative disorders (PTLD) associated lymphomas.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- United States (8):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Johns Hopkins Oncology Center ORA, Baltimore, Maryland
  - Dana Farber Cancer Institute Dept.of DFCI, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center MSKCC (8), New York, New York
  - Cinn Children Hosp Medical Center, Cincinnati, Ohio
  - The Childrens Hospital of Philadelphia Drug Shipment, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center ., Dallas, Texas
- Australia (2):
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Helsinki, Finland
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Münster, Germany
- Italy (2):
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Roma, RM
- Japan (2):
  - Kyoto University Hospital, Sakyō-ku, Kyoto
  - Novartis Investigative Site, Setagaya-ku, Tokyo
- Prinses Maxima Centrum voor Kinderoncologie, Utrecht, CS, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in twenty-four centers across 14 countries. Although 34 participants met the eligibility criteria and apheresis was accepted by the manufacturing facility, only 33 were infused in the study.
Pre-assignment Details: Consent, Screening, Pre-treatment, Treatment and Follow-up. In the Pretreatment phase, the subject may have undergone optional bridging therapy or lymphodepleting chemotherapy. Full Analysis Set: 33 Efficacy Analysis Set (EAS): 28; 4 patients with Complete Response prior to infusion & 1 without a scan prior to infusion excluded from EAS.
Groups:
- Tisagenlecleucel: These participants were infused once with CAR-positive viable T cells.
Period: Overall Study
Arm/Group | Tisagenlecleucel
Started | 34
Met Eligibilty Criteria and Were Infused | 33
Met Eligibilty Criteria But Was Not Infused* (*Patient died prior to infusion) | 1
Completed Treatment & Primary Follow-up Phase | 14
Discont. Treatment & Primary Follow-up Phase | 19
Completed | 14
Not Completed | 20
Not completed — Death | 17
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Died prior to infusion | 1

BASELINE CHARACTERISTICS:
Population: FAS and safety set: all subjects who received an infusion of tisagenlecleucel
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 33
Age, Continuous [Median (Standard Deviation); unit: years] | 12.8 (4.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 23
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 28
  Black or African American | 1
  Asian | 2
  Missing | 2
Histology (type of lymphoma) [Count of Participants; unit: Participants]
  Burkitt lymphoma | 18
  Large B-cell lymphoma | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Determined by Local Investigator
Description: The overall response rate (ORR) is defined as the percentage of subjects with a best overall disease response of complete response (CR) or partial response (PR), where the best overall disease response is defined as the best disease response recorded from tisagenlecleucel infusion until progressive disease or start of new anticancer therapy, whichever comes first.
Time Frame: 6 months post-tisagenlecleucel infusion
Population: Efficacy Analysis Set (EAS): all subjects with aggressive r/r B-cell NHL who received an infusion of tisagenlecleucel and had measurable disease at baseline, i.e participants with complete or unknown response after bridging therapy were excluded from the efficacy analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 28
Percentage of participants | 32.1 [15.9 to 52.4]

2. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) is defined as the time from the date of first documented disease response (CR or PR) as determined by local investigator assessments to the date of first documented progression or death due to underlying cancer.
Time Frame: Post-infusion Day 28, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24, and then annually until Month 48
Population: EAS: all subjects with aggressive r/r B-cell NHL who received an infusion of tisagenlecleucel and had measurable disease at baseline. Only participants with best response of CR/PR post-infusion were included in the DOR analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 9
months | NA [1.0 to NA] — NA: Median and Upper limit of Confidence Interval (CI) not reached because there were not sufficient events during study follow-up

3. Secondary Outcome: Event Free Survival (EFS)
Description: Event free survival (EFS) is defined as the time from date of first tisagenlecleucel infusion to the earliest date of death from any cause, disease progression as determined by local investigator assessments, or starting new anticancer therapy for underlying cancer, excluding hematopoietic stem cell transplant (HSCT).
Time Frame: Post-infusion Day 28, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24, and then annually until Month 48
Population: EAS: all subjects with aggressive r/r B-cell NHL who received an infusion of tisagenlecleucel and had measurable disease at baseline, i.e participants with complete or unknown response after bridging therapy were excluded from the efficacy analysis set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 28
months | 2.1 [1.1 to 2.8]

4. Secondary Outcome: Relapse Free Survival (RFS)
Description: Relapse free survival (RFS) is defined as the time from the date of first documented disease response (CR or PR) as determined by local investigator assessments to the date of first documented disease progression or death due to any cause.
Time Frame: Post-infusion Day 28, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24, and then annually until Month 48
Population: EAS: all subjects with aggressive r/r B-cell NHL who received an infusion of tisagenlecleucel and had measurable disease at baseline. Only participants with best response of CR/PR post-infusion were included in the RFS analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 9
months | NA [1.0 to NA] — NA: Median and Upper limit of Confidence Interval (CI) not reached because there were not sufficient events during study follow-up

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from the date of first tisagenlecleucel infusion to the date of first documented disease progression as determined by local investigator assessments or death due to any cause.
  Progression is defined using the International non-Hodgkin Lymphoma Response Criteria. For a PET-based response, progressive disease is defined as a 4 or 5 on the 5 point scale with increased uptake compared to the nadir or new FDG-avid foci consistent with lymphoma. For a CT/MRI based response progressive disease is defined as a 25% increase in the SPD (sum of the products of two largest perpendicular diameters) of index lesions, or unequivocal progression in either non-index lesions or the spleen. Any new disease attributable to lymphoma would also constitute progressive disease.
Time Frame: Post-infusion Day 28, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24, and then annually until Month 48
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 28
months | 2.5 [1.1 to 2.9]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from date of first tisagenlecleucel infusion to the date of death due to any cause.
Time Frame: Post-infusion Day 28, Month 3, Month 6, Month 9, Month 12, Month 18, Month 24, and then annually until Month 48
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 28
months | 10.4 [3.4 to NA] — NA: Upper limit of Confidence Interval (CI) not reached because there were not sufficient events during study follow-up

7. Secondary Outcome: Cellular Kinetics Parameter: Cmax
Description: The maximum (peak) transgene level (copies/μg) observed in peripheral blood or other body fluid after single dose administration as measured by qPCR. Pharmacokinetics of tisagenlecleucel were based on chimeric antigen receptor (CAR) transgene levels in peripheral blood as detected by qPCR, unless otherwise noted. Pharmacokinetics of tisagenlecleucel were based on chimeric antigen receptor (CAR) transgene levels in peripheral blood as detected by qPCR, unless otherwise noted.
Time Frame: Post-infusion day 4, day 7, day 11, day 14, day 21, day 28, month 3, month 6, month 9, month 12, month 18, month 24, and then annually until Month 48
Population: Cellular kinetic analysis set (CKAS): subjects in the FAS who provided at least 1 valid cellular kinetic concentration for tisagenlecleucel. Certain PK parameters were not estimable for all subjects due to insufficient samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/μg
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 31
copies/μg | 5140 (238.9)

8. Secondary Outcome: Cellular Kinetics Parameter: Tmax
Description: The time to reach maximum (peak) transgene level (days) in peripheral blood or other body fluid after single dose administration. Pharmacokinetics of tisagenlecleucel were based on chimeric antigen receptor (CAR) transgene levels in peripheral blood as detected by qPCR, unless otherwise noted.
Time Frame: as for outcome 7
Population: CKAS: subjects in the FAS who provided at least 1 valid cellular kinetic concentration for tisagenlecleucel. Certain PK parameters were not estimable for all subjects due to insufficient samples.
Measure: Median (Full Range); unit: days
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 31
days | 12.7 [1.90 to 21.9]

9. Secondary Outcome: Cellular Kinetics Parameter: AUC0-28d
Description: Area Under the Concentration-time Curve (AUCs) from the time course of transgene levels in peripheral blood following tisagenlecleucel infusion (days*copies/μg), from day of infusion to day 28. D28 refers to the timepoint for definition of responder populations. Pharmacokinetics of tisagenlecleucel were based on chimeric antigen receptor (CAR) transgene levels in peripheral blood as detected by qPCR, unless otherwise noted.
Time Frame: 0 to 28 days
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/μg*days
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 27
copies/μg*days | 53500 (154.9)

10. Secondary Outcome: Cellular Kinetics Parameter: Clast
Description: The last observed quantifiable transgene level in peripheral blood. Pharmacokinetics of tisagenlecleucel were based on chimeric antigen receptor (CAR) transgene levels in peripheral blood as detected by qPCR, unless otherwise noted.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: copies/μg
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 30
copies/μg | 344 (350.4)

11. Secondary Outcome: Cellular Kinetics Parameter: Tlast
Description: The time of last observed quantifiable transgene level in peripheral blood. Pharmacokinetics of tisagenlecleucel were based on chimeric antigen receptor (CAR) transgene levels in peripheral blood as detected by qPCR, unless otherwise noted.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Median (Full Range); unit: days
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 30
days | 40.0 [13.0 to 1090]

12. Secondary Outcome: Levels of Pre-existing and Treatment Induced Humoral Immunogenicity and Cellular Immunogenicity Against Tisagenlecleucel Cellular Kinetics, Safety and Efficacy
Description: The humoral immunogenicity assay measures the antibody titers specific to tisagenlecleucel prior to and following infusion by flow cytometry. A subject was only defined as positive for tisagenlecleucel treatment-induced or -boosted anti-mCAR19 antibodies when the anti-mCAR19 antibody median fluorescence intensity at any time post-infusion was at least 2.28-fold higher (for samples analyzed on or prior to 05-May-2021) or 2.38-fold higher (for samples analyzed on or after 06-May-2021) than pre-infusion levels for participants whose baseline status was positive (boosted) or if the baseline status was negative but any post-baseline interpretation was positive (induced).
Time Frame: Until disease progression or through study completion, up to 4 years
Population: Safety set: All participants who received an infusion of tisagenlecleucel
Measure: Number; unit: Percentage of participants
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 33
Percentage of participants
  anti-tisagenlecleucel antibodies (positive) at baseline (BL) | 87.9
  anti-tisagenlecleucel antibodies (positive) anytime post-BL | 97.0

13. Secondary Outcome: Percentage of Participants Who Proceeded to Stem Cell Transplant (SCT) After Tisagenlecleucel Infusion
Description: These participants proceeded to transplant any time post-tisagenlecleucel therapy until end of study (EOS).
Time Frame: Through study completion, up to 4 years
Population: Safety set: All participants who received an infusion of tisagenlecleucel
Measure: Number; unit: Percentage of participants
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 33
Percentage of participants | 21.2 [9.0 to 38.9]

14. Secondary Outcome: Maximum Positive Predictive Value (PPV)
Description: Retrospective assessment of potential cytokine release syndrome (CRS) predictive models considering also data from other CTL019 trials. The Positive Predictive Value (PVV) is the percentage of participants who actually had severe CRS out of all the cases where the prediction model predicts that severe CRS will occur. The maximum PPV is the highest value attained across all potential CRS predictive models.
Time Frame: Through study completion, up to 4 years
Population: Safety set: All participants who received an infusion of tisagenlecleucel
Measure: Number; unit: Percentage of participants
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 33
Percentage of participants | 36.0

15. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected during the post-infusion period starting at the day of first infusion until the end of the study, up to 48 months. All deaths is the sum of pre-infusion and post-infusion deaths.
Time Frame: Pre-treatment deaths: from enrollment to pre-infusion; On-treatment deaths: post-infusion up to 48 months
Population: Clinical Database Population: All infused and non-infused participants who met the criteria to be enrolled in the study
Measure: Number; unit: Participants
Arm/Group | Tisagenlecleucel
Number analyzed (Participants) | 34
Participants
  On-treatment deaths include post-treatment survival follow-up deaths | 17
  Deaths prior to infusion | 1
  All Deaths | 18

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) timeframe: AEs were collected during the post-infusion period (starting at the day of 1st infusion until the end of the study), up to maximum duration of 48 months for each patient. Deaths were collected at all points: pre-infusion period and post-infusion period until the patient completed the study duration (48 months) or further safety follow-up under the study protocol. Therefore on-treatment deaths include post-infusion deaths until Last patient Last Visit (LPLV)
Description: AE description: Any sign or symptom that occurs during the post-infusion period (starting at the day of first infusion of CTL019 until the end of the study) and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events while still included in the All-Cause Mortality table.
Groups:
- Tisagenlecleucel - Post-infusion: AEs/deaths collected during and post- infusion until patient completed study.
- Tisagenlecleucel - Pre-infusion Deaths: Deaths collected prior to infusion. No AEs were collected during this period.
Arm/Group | Tisagenlecleucel - Post-infusion | Tisagenlecleucel - Pre-infusion Deaths
All-Cause Mortality (participants affected / at risk) | 17/33 | 1/34
Serious Adverse Events (participants affected / at risk) | 24/33 | 0/0
Other Adverse Events (participants affected / at risk) | 33/33 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel - Post-infusion (N=33) | Tisagenlecleucel - Pre-infusion Deaths (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | NA
Cardiac arrest (Cardiac disorders) | 1 | NA
Tachycardia (Cardiac disorders) | 1 | NA
Vision blurred (Eye disorders) | 1 | NA
Abdominal pain (Gastrointestinal disorders) | 2 | NA
Dental caries (Gastrointestinal disorders) | 1 | NA
Large intestinal obstruction (Gastrointestinal disorders) | 1 | NA
Pancreatitis (Gastrointestinal disorders) | 1 | NA
Proctitis (Gastrointestinal disorders) | 1 | NA
Chest pain (General disorders) | 1 | NA
Condition aggravated (General disorders) | 1 | NA
Disease progression (General disorders) | 1 | NA
Pyrexia (General disorders) | 7 | NA
Cytokine release syndrome (Immune system disorders) | 8 | NA
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | NA
Aspergillus infection (Infections and infestations) | 1 | NA
Candida infection (Infections and infestations) | 1 | NA
Pseudomonas infection (Infections and infestations) | 1 | NA
Sepsis (Infections and infestations) | 1 | NA
Urinary tract infection (Infections and infestations) | 1 | NA
Vascular device infection (Infections and infestations) | 1 | NA
Ejection fraction decreased (Investigations) | 1 | NA
Neutrophil count decreased (Investigations) | 1 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | NA
Aphasia (Nervous system disorders) | 1 | NA
Depressed level of consciousness (Nervous system disorders) | 2 | NA
Disturbance in attention (Nervous system disorders) | 1 | NA
Hemiparesis (Nervous system disorders) | 1 | NA
Memory impairment (Nervous system disorders) | 1 | NA
Motor dysfunction (Nervous system disorders) | 1 | NA
Peripheral sensorimotor neuropathy (Nervous system disorders) | 2 | NA
Seizure (Nervous system disorders) | 2 | NA
Acute kidney injury (Renal and urinary disorders) | 2 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Hypertension (Vascular disorders) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel - Post-infusion (N=33) | Tisagenlecleucel - Pre-infusion Deaths (N=0)
Anaemia (Blood and lymphatic system disorders) | 11 | NA
Bone marrow failure (Blood and lymphatic system disorders) | 2 | NA
Coagulopathy (Blood and lymphatic system disorders) | 2 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | NA
Leukopenia (Blood and lymphatic system disorders) | 5 | NA
Lymphopenia (Blood and lymphatic system disorders) | 2 | NA
Neutropenia (Blood and lymphatic system disorders) | 7 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | NA
Sinus tachycardia (Cardiac disorders) | 3 | NA
Tachycardia (Cardiac disorders) | 4 | NA
Vision blurred (Eye disorders) | 2 | NA
Abdominal pain (Gastrointestinal disorders) | 6 | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 | NA
Constipation (Gastrointestinal disorders) | 3 | NA
Diarrhoea (Gastrointestinal disorders) | 3 | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | NA
Nausea (Gastrointestinal disorders) | 9 | NA
Small intestinal obstruction (Gastrointestinal disorders) | 2 | NA
Stomatitis (Gastrointestinal disorders) | 5 | NA
Vomiting (Gastrointestinal disorders) | 13 | NA
Catheter site pain (General disorders) | 3 | NA
Chills (General disorders) | 4 | NA
Fatigue (General disorders) | 5 | NA
Generalised oedema (General disorders) | 2 | NA
Oedema peripheral (General disorders) | 2 | NA
Pain (General disorders) | 2 | NA
Pyrexia (General disorders) | 14 | NA
Cholelithiasis (Hepatobiliary disorders) | 2 | NA
Cytokine release syndrome (Immune system disorders) | 16 | NA
Drug hypersensitivity (Immune system disorders) | 2 | NA
Hypogammaglobulinaemia (Immune system disorders) | 3 | NA
Myelitis (Infections and infestations) | 2 | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | NA
Alanine aminotransferase increased (Investigations) | 5 | NA
Aspartate aminotransferase increased (Investigations) | 2 | NA
Blood bilirubin increased (Investigations) | 2 | NA
Blood creatinine increased (Investigations) | 5 | NA
Blood lactate dehydrogenase increased (Investigations) | 3 | NA
Lymphocyte count decreased (Investigations) | 3 | NA
Neutrophil count decreased (Investigations) | 10 | NA
Platelet count decreased (Investigations) | 9 | NA
SARS-CoV-2 test positive (Investigations) | 2 | NA
Serum ferritin increased (Investigations) | 2 | NA
Weight decreased (Investigations) | 3 | NA
White blood cell count decreased (Investigations) | 8 | NA
Decreased appetite (Metabolism and nutrition disorders) | 5 | NA
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 5 | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | NA
Depressed level of consciousness (Nervous system disorders) | 2 | NA
Dizziness (Nervous system disorders) | 2 | NA
Headache (Nervous system disorders) | 8 | NA
Neuralgia (Nervous system disorders) | 2 | NA
Neuropathy peripheral (Nervous system disorders) | 2 | NA
Paraesthesia (Nervous system disorders) | 3 | NA
Anxiety (Psychiatric disorders) | 2 | NA
Depression (Psychiatric disorders) | 2 | NA
Insomnia (Psychiatric disorders) | 2 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Alopecia (Skin and subcutaneous tissue disorders) | 2 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 2 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 | NA
Rash (Skin and subcutaneous tissue disorders) | 2 | NA
Haematoma (Vascular disorders) | 2 | NA
Hypertension (Vascular disorders) | 3 | NA
Hypotension (Vascular disorders) | 2 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03610724/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT03610724/SAP_001.pdf